CLINICAL TRIAL: NCT06110312
Title: Study Protocol for an International Pragmatic Randomised Controlled Trial of the NavCare-EU Intervention for Older People With Cancer and Their Family Caregivers
Brief Title: International Study to Evaluate a Navigation Program for Older People With Cancer and Their Family Caregivers (EU NAVIGATE Study)
Acronym: EU NAVIGATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University of Dublin, Trinity College (Other); Uniwersytet Jagiellonski (Unknown); Amsterdam UMC, location VUmc (Other); University of Coimbra (Other); University Ghent (Other); University of British Columbia (Other); Lega Italiana per la Lotta contro i Tumori (Other)
Responsible Party: Principal Investigator, Lieve Van den Block, Professor of ageing and palliative care, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1432023000143; 101057361 (Other Grant/Funding Number: Horizon Europe)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Cancer (Active Cancer, Meaning Not Being Cancer Free), of Any Stage and Involving Any Treatment/Care Regimen; i.e. Curative, Life-extending, or Palliative
Keywords: palliative care; supportive care; cancer; family caregiver; older people; community; primary care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In EU NAVIGATE, participants in the intervention group will receive a navigation intervention (also called NavCare-EU), alongside any usual care. Navcare-EU is a person- and family-centered navigation intervention, aimed at supporting older people with cancer throughout the care and illness continuum, via the involvement of a patient/family navigator. Navigators focus on connecting clients to social supports, both formal and informal, advocating for clients in meeting their quality-of-life goals, resourcing by identifying needs and negotiating access to meeting those needs, and engaging clients in what is most meaningful to them. Navigators are selected, trained, and mentored volunteers or professionals. NavCare-EU is based on the existing and successfully tested Nav-CARE(c) intervention from Canada.
  Interventions: Behavioral: NavCare-EU
- control group (No Intervention): Participants in the control group will receive what is usual care in each of the participating countries for 24 weeks (primary trial outcome). After 24 weeks, they will also receive the navigation intervention (NavCare-EU) (fast-track RCT).

INTERVENTIONS:
Behavioral: NavCare-EU — NavCare-EU is a person- and family-centered intervention in which navigators collaborate with older persons and their close family caregivers across the continuum of supportive, palliative, and end-of-life care,. NavCare-EU is based on the existing and successfully tested Nav-CARE intervention from Canada. Navigators focus on connecting clients to social supports, both formal and informal, advocating for clients in meeting their quality-of-life goals, resourcing by identifying needs and negotiating access to meeting those needs, and engaging clients in what is most meaningful to them. Navigators are selected, trained, and mentored volunteers or professionals. NavCare-EU is based on the existing and successfully tested Nav-CARE(c) intervention from Canada.
  Arms: intervention group

SUMMARY:
Most people with cancer are older, and this affects millions of Europeans yearly. Integrating high-quality, equitable, and cost-effective care across the continuum of supportive, palliative, and end-of-life care for both patients and family caregivers is highly relevant from a healthcare, prevention, and economic perspective.

EU NAVIGATE is an interdisciplinary, cross-country, and intersectoral project funded by the European Union. The overall aim of the study is to evaluate the effectiveness and cost-effectiveness of a patient and family navigation intervention (NavCare-EU) for older people with cancer and declining health and their family caregivers in different healthcare systems in Europe. Nav-Care EU is a person- and family-centered non-pharmacological intervention in which navigators collaborate with patients and families to improve quality of life and improve levels of social support, foster empowerment, and facilitate timely and equitable access to health and social care services and resources as needed, throughout the supportive and palliative care continuum. NavCare-EU is based on the existing and successfully tested Nav-CARE(c) intervention from Canada.

Effectiveness and cost-effectiveness will be evaluated through an international 6-country multisite pragmatic fast-track randomised controlled trial (RCT) with an embedded mixed methods process evaluation to compare the NavCare-EU intervention in addition to standard care with the provision of standard care alone. The RCT and process evaluation will be conducted in Belgium (Flanders), Ireland, Italy, the Netherlands, Poland, and Portugal. Participants are people with cancer and declining health, who are aged 70 years and older, as well as their close family caregivers.

Specific objectives are:

1. To compare the NavCare-EU intervention to care as usual, in terms of its:

1. Effectiveness on (1) global health status/quality of life, and the levels of social support (two co-primary outcomes); and on feelings of loneliness of older persons with cancer across the continuum of supportive, palliative, and end-of-life care; (2) family caregiver burden
2. cost-effectiveness
3. effects on different subgroups defined by characteristics known to affect health equity and equitable access, i.e., gender, age, socioeconomic status, extent of social support and living situation, and geographical location (rural vs. urban)
4. effectiveness and cost-effectiveness in different health care systems and care regimes in Europe

2. To evaluate the implementation processes of the NavCare-EU intervention and the feasibility of its integration in different health care systems and care regimens in Europe, the contextual barriers and facilitators for effective and sustainable implementation, and the mechanisms involved in reaching the outcomes in each country, as perceived by patients, family caregivers, and other care providers

ELIGIBILITY:
For older person with cancer

Inclusion criteria

* Have a cancer diagnosis (active cancer, meaning not being cancer free, of any stage and involving any treatment/care regimen; i.e. curative, life-extending, or palliative), AND
* Aged 70 years or over, AND
* Have declining or deteriorating health using the Clinical Frailty Scale, AND
* Live at home (own home or home of the family caregiver) (or discharged home if recruited in hospital), AND
* Live within the catchment area of the navigation programme/service

Exclusion criteria

* The close family caregiver living with the person with cancer or providing care at least on a weekly basis, and identified as the primary family caregiver by the person with cancer, if present, does not agree to participate in the study (unless participation is explicitly requested by the patient) , OR
* Lives in a care or nursing home, or is incarcerated, OR
* Currently receives care from a formally recognized community-based multidisciplinary or specialist palliative care team, OR
* Is unable to provide informed consent or has difficulties understanding the information about the study , OR
* Has a psychiatric condition (i.e. schizophrenia, bipolar disorder, or major depressive disorder) OR has an active substance abuse disorder OR
* Is not able to participate in data collection in the country's language

For close family caregiver (if present)

Inclusion criteria

* Aged 18 years or over , AND
* Lives with the person with cancer OR provides care at least on a weekly basis, AND
* Identified as primary family caregiver by the older person with cancer

Exclusion criteria

* Is unable to provide informed consent or has difficulties understanding the information about the study, OR
* Is not able to participate in data collection in the country's language

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 489 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Global health status/quality of life of the older person with cancer | Change from baseline at 24 weeks.
  Global health status/quality of life of the older person with cancer, measured with 2-item subscale from the EORTC-QLQ-C30 (revised) measuring health-related quality of life.
Levels of social support of the older person with cancer | Change from baseline at 24 weeks.
  Levels of social support of the older person with cancer measured with the Medical Outcomes Study Social Support Survey (MOS)

SECONDARY OUTCOMES:
Feelings of loneliness of the older person with cancer | Change from baseline at 24 weeks.
  Feelings of loneliness (relational and social connectedness, and self-perceived isolation) of the older person with cancer, measured with the 3-item-UCLA Revised Loneliness Scale.
Caregiver burden of close family caregivers | Change from baseline at 24 weeks.
  Caregiver burden of close family caregivers, measured with the Zarit Burden Interview Short Form

OTHER OUTCOMES:
Global health status/quality of life of the older person with cancer | Change from baseline at 48 weeks.
  Global health status/quality of life of the older person with cancer, measured with 2-item subscale from the EORTC-QLQ-C30 (revised) measuring health-related quality of life.
Levels of social support of the older person with cancer | Change from baseline at 48 weeks.
  Levels of social support of the older person with cancer measured with the Medical Outcomes Study Social Support Survey (MOS)
Feelings of loneliness of the older person with cancer | Change from baseline at 48 weeks.
  Feelings of loneliness (relational and social connectedness, and self-perceived isolation) of the older person with cancer, measured with the 3-item-UCLA Revised Loneliness Scale.
Caregiver burden of close family caregivers | Change from baseline at 48 weeks.
  Caregiver burden of close family caregivers, measured with the Zarit Burden Interview Short Form
Symptoms or problems experienced | Change from baseline at 24 weeks.
  Symptoms or problems experienced (i.e. as measured by the EORTC-QLQ-C30 symptom subscales and the emotional functioning scale for cancer patients
well-being of older people | Change from baseline at 24 weeks.
  well-being of older people (WOOP) (which captures a comprehensive set of well-being domains relevant to older people (broader than health)
Knowledge of resources and services and confidence in decision making and communicating those decisions | Change from baseline at 24 weeks.
  Knowledge of resources and services and confidence in decision making and communicating those decisions (measured with the Nav-CARE engagement questionnaire).
Health status | Change from baseline at 24 weeks.
  Health status EQ-5D (has traditionally been used as outcome measure in economic evaluations)
Health and social care services and resource use | Change from baseline at 24 weeks.
  Health and social care services and resource use (for economic evaluation)
positive aspects of caregiving of close family caregivers (measured with PAC scale) | Change from baseline at 24 weeks.
  positive aspects of caregiving of close family caregivers (measured with PAC scale)

CONTACTS AND LOCATIONS:
Overall Officials: Lieve Van den Block, PhD, Principal Investigator — Vrije Universiteit Brussel

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be made available to third parties upon reasonable request and upon signing a unilateral data sharing agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: The data can be obtained from the authors of the publication upon reasonable request. Data will be shared with members of universities, scientific research institutions, or clearly separate and independent research departments of public institutions or non- profit organisations. Data may be used for scientific research only (commercial use of data will not be permitted).

REFERENCES:
- [Derived] Smets T, Pivodic L, Miranda R, Van Campe F, Vinckier C, Pesut B, Duggleby W, Davies AN, Lavan A, May P, Gomes B, Furlan de Brito M, Rodrigues V, Szczerbinska K, Kijowska V, Baranska I, De Buyser S, Ferraris D, Alfieri S, Scacciati B, Du Cheyne H, Chambaere K, Gilissen J, van der Plas AGM, Pasman RH, Onwuteaka-Philipsen BD; EU NAVIGATE; Van den Block L. Implementation and evaluation of a navigation program for people with cancer in old age and their family caregivers: study protocol for the EU NAVIGATE International Pragmatic Randomized Controlled Trial. Trials. 2024 Nov 27;25(1):800. doi: 10.1186/s13063-024-08633-5. PMID 39605055